CLINICAL TRIAL: NCT01864460
Title: Improving Autonomic Function and Balance in Diabetic Neuropathy
Acronym: IMABIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E1030-R
Record Dates: First submitted 2013-05-16; First posted 2013-05-29 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Diabetes; Neuropathy; Impaired Glucose Tolerance
Keywords: autonomic; neuropathy; balance; exercise
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diet, Physical Activity and Balance Enhancement Program (DPAE (Experimental): Subjects in the DPAEP group will undergo a structured weight loss for approximately 6 months, followed by approximately 6 months of weight maintenance, as well as 12 months of aerobic exercise. This intervention stresses a personalized program emphasizing activities that are meaningful to and are tailored to individual participants; provides consistent contact between the participants and research staff; and allows monitoring of activity levels using questionnaires, actigraphy, monitoring of heart rate, direct and telephone contact. Participants dietary and physical activity goals as assessed by the dietician and trainer will be discussed at face-to face meetings to re-establish these goals. These programs will be tailored to meet the realistic goals of the individual participant. The program stresses aerobic exercise, rather than other types of exercise interventions, as aerobic exercise appears to correlate best with improved autonomic function.
  Interventions: Behavioral: lifestyle modification
- Standard Care (SC) (Active Comparator): The SC group will be assigned an interventionist assessor. This assessor will meet with the subjects during their orientation meeting and will be provided guidelines and a weight loss and physical activity target to achieve by the end of the program at their orientation meeting. Participants will contacted approximately weekly during the approximate 12 month period.
  Interventions: Behavioral: lifestyle modification

INTERVENTIONS:
Behavioral: lifestyle modification — Structured weight loss or weight maintenance and aerobic exercise intervention for 12 months or standard of care weight and exercise management

SUMMARY:
Type 2 diabetes (DM2) affects nearly 20 million people in the United States while impaired glucose regulation (IGR), which includes impaired glucose tolerance (IGT), impaired fasting glucose (IFG), and early diabetes affects a considerably larger but unknown population group. At the current time there is no effective therapy to completely prevent, or reverse neuropathy associated with IGR and this represents a considerable challenge in rehabilitation. There is a particularly strong incentive to prevent IGT and related complications from advancing to DM2. IGR is a growing problem among all older adults and its strong association with many functional limitations, particularly mobility limitations, is not always recognized, even though diabetes-related disability occurs in up to 2/3 of older adults with diabetes and is associated with dependency, poor quality of life, and increased acute and long-term care utilization.

Autonomic dysfunction is a significant problem in subjects with IGT. The Preliminary Data shows that over 90% of subjects with IGT have an abnormal score on questionnaires about autonomic symptoms such as lightheadedness, dry mouth or dry eyes, pale or blue feet, feet that are colder than the rest of the body, decreased sweating in the feet or increased sweating in the hands, nausea or bloating after eating, persistent diarrhea or constipation, or leaking of urine. In addition, patients with IGR have impaired balance control. These factors can increase the risk of falls in affected subjects. A non-randomized and non-controlled study showed that a diet and exercise intervention in patients with diabetes led to an overall improvement in autonomic function. Furthermore, it was shown that standing balance can be improved with a balance intervention program.

However, there are no published studies that assess the effect of an intense physical activity intervention on autonomic function in IGR related neuropathy. This study will test an aerobic exercise and balance intervention in participants with IGR. The investigators will examine if an individually tailored, carefully monitored, Diet, Physical Activity, and Balance Enhancement Program (DPAEP) can improve autonomic function and balance control when compared to patients who receive standard care. Improving balance control and autonomic function can decrease the risk of falls and have a significant effect on the health of participants.

The research is also significant because it will test subjects either before they become diabetic, or at an early stage in their diabetes, thus enhancing the chance of reversing the autonomic neuropathy or balance impairment. Furthermore, the study is designed to test whether improvement in autonomic function and balance is associated with improvement in clinical outcomes, quality of life, and the metabolic state of participants. Thus, the proposed interventions are likely to have a real life impact on participants and their health.

DETAILED DESCRIPTION:
Study on hold due to COVID-19

In this proposed study, investigators will determine if an intense, individually tailored, carefully monitored, Diet, Physical Activity and Balance Enhancement Program (DPAEP) can improve autonomic function and balance and other measures of autonomic and balance control. In contrast, the primary and secondary and other efficacy measures will be compared in standard care controls (SC) who will receive general diet and physical activity information. The "Improving Autonomic Function and Balance in Diabetic Neuropathy" study is a single blinded, randomized study to determine if an intensive diet and exercise program improves autonomic function and balance. Following baseline testing, participants are randomized to either DPAEP or SC groups. DPAEP participants will receive an intensive physical activity enhancement program with a focus on aerobic activity and a balance program.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose regulation at the time of screening or within three months of screening. This definition includes patients with IFG, IGT, and early or mild DM2. Patients can be included if they have an increased risk for diabetes with a HBA1C greater than or equal to 5.7% (using a method certified by the National Glycohemoglobin Standardization Program), or they have diabetes with a HBA1C greater than or equal to 6.5%, or an abnormal fasting venous glucose, or abnormal venous glucose values following a 75 gram oral glucose load. Glucose values are as defined (mg/dl): IFG fasting glucose of 100-125 mg/dl, IGT- fasting less than 126, 2 h 140-199, or diabetes - fasting glucose greater than or equal to 126, or 2 h greater than or equal to 200 based on the Standards for Medical Care in Diabetes 2010 by the American Diabetes Association.
* The HbA1c may be normal, but should be less than 9%.
* If diabetic subjects are on medication, they should be stable on medication for at least 3 months prior to entering the study. Addition or change in antidiabetic medication (if on medication) after enrollment does not affect participation or group assignment.
* Impaired glucose regulation is the most likely cause of the neuropathy (determined by a medical history, family history, history of medications, occupational history, history of exposure to toxins (including significant alcohol use), physical and neurological examinations, and appropriate laboratory studies.
* Autonomic neuropathy as defined by the Toronto Diabetic Neuropathy Expert Group 2010/11 consensus criteria. Subjects with be entered into the study if they have (1) increased symptoms of autonomic neuropathy based on an increase in the number of symptoms (>3) OR impact score (>7) in the validated SAS OR (2) at least two abnormalities on autonomic testing. The autonomic testing includes: (a) heart rate variability (E:I ratio and heart rate range-HRR), (b) Valsalva ratio, (c) Valsalva beat to beat blood pressure variation, (d) 30:15 ratio, (e) tilt table testing, and (f) QSART values.
* Age 30 (to exclude patients with type 1 diabetes) to 80 years inclusive
* Medically stable at the time of enrollment.
* Women of childbearing potential must be using an acceptable method of contraception to prevent pregnancy when they are enrolled in the study and must agree to continue to practice an acceptable method of contraception for the duration of their participation in the study.
* Patient must agree to take an alternative medication to coumadin when undergoing a skin biopsy.

Exclusion Criteria:

* Pregnant women, prisoners, institutionalized subjects and other at risk subjects will not be included in this study.
* Neuropathy due to factors other than impaired glucose regulation based on careful clinical and laboratory evaluation by the physician.
* Current severe medical conditions that are active on the day of screening that would affect the patient's ability to participate in or complete the study.
* Autonomic neuropathy that is so severe that it would limit the patient's ability to participate in the study interventions.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11-14 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Autonomic Function: heart rate variability | 12 months
  This is a cardiac autonomic measure that will be carried out using clinical equipment in the autonomic laboratory at the site. The measurement requires placing electrodes near the heart similar to an EKG.

SECONDARY OUTCOMES:
balance | 6 and 12 months
  This outcome measure assesses changes in trunk positioning using a standardized, validated test.

OTHER OUTCOMES:
Sweat gland nerve fiber density | 12 months
  This outcome assesses sweat gland nerve fiber density, which is proposed as a sensitive neuropathy pathology biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: James W Russell, MD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No